CLINICAL TRIAL: NCT04371107
Title: Proactive Care of Ambulatory COVID19 Patients: Open-labeled Randomized Trial
Brief Title: Proactive Care of Ambulatory COVID19 Patients
Acronym: AMBU-COVID
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: ANSM notifications
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2020_843_0039
Record Dates: First submitted 2020-04-27; First posted 2020-05-01 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Azithromycin; Ambulatory
Keywords: Covid19; azithromycine; ambulatory
MeSH Terms: conditions — COVID-19 | interventions — Referral and Consultation; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- azithromycin (Experimental): azithromycin treatment 500 mg on day 1 then 250 mg the following 4 days from day 2 to day 5, per os.
  Interventions: Other: consultation; Drug: Azithromycin
- symptomatic treatment (Active Comparator): continuation of symptomatic treatment
  Interventions: Other: consultation

INTERVENTIONS:
Other: consultation — Patients are followed up by teleconsultation or remote follow-up until the end of symptoms and for a maximum of 2 months
Drug: Azithromycin — azithromycin treatment 500 mg on day 1 then 250 mg the following 4 days from day 2 to day 5, per os.
  Arms: azithromycin

SUMMARY:
On January 9, 2020, a new emerging virus was identified by WHO as being responsible for grouped cases of pneumonia in China. It is a coronavirus, SARS-CoV-2, responsible for the disease COVID-19 (Coronavirus disease). The disease is mild in 85% of cases but the proportion of serious cases requiring hospitalization or intensive care (15%) puts stress on health structures and systems around the world.

To limit the influx of patients and avoid overstretching Health systems, containment and social distancing strategies are widely adopted.

It appears crucial to propose the easiest possible therapeutic strategy taking into account the ambulatory nature of the patients. Therefore azithromycin (AZM) is an antibiotic known to have an antiviral effect but also which has anti-inflammatory activity in addition to its antimicrobial effect. Azithromycin targets preferentially pulmonary cells (and particularly of the lines apparently affected in COVID-19 positive cases). The aim of this study is to demonstrate that AZM decreases symptom duration in COVID19 patients and diminishes the viral carriage.

DETAILED DESCRIPTION:
On January 9, 2020, a new emerging virus was identified by WHO as being responsible for grouped cases of pneumonia in China. It is a coronavirus, SARS-CoV-2, responsible for the disease COVID-19 (Coronavirus disease). The disease is mild in 85% of cases but the proportion of serious cases requiring hospitalization or intensive care (15%) puts stress on health structures and systems around the world.

To limit the influx of patients and avoid overstretching Health systems, containment and social distancing strategies are widely adopted.

It appears crucial to propose the easiest possible therapeutic strategy taking into account the ambulatory nature of the patients. Treatment must be as safe as possible allowing a wide distribution to the symptomatic population while keeping a favorable risk/benefice balance for a patient with little symptoms.

Several studies show that azithromycin (AZM) has an anti-inflammatory effect. In patients with cystic fibrosis, AZM is known to have an anti-fibrotic effect by targeting myofibroblast cells, which considerably prolongs their lifespan. AZM acts functionally as an anti-inflammatory drug and reduces senescence associated secretory phenotype (SASP) mediators, such as IL-1beta and IL-632. AZM has also been shown to inhibit the replication of certain viruses, such as Zika and Ebola.

Therefore AZM is an antibiotic known to have an antiviral effect but also which has anti-inflammatory activity in addition to its antimicrobial effect. Azithromycin targets preferentially pulmonary cells (and particularly of the lines apparently affected in COVID-19 positive cases) Therefore, the prescription of AZM in COVID-19 + patients aims to increase the antiviral response locally at pulmonary level, while promoting a decrease in the immune response at systemic level.

Its specific effect and excellent clinical tolerance justifies its use as monotherapy in non-severe covid-19 + cases for the present study.

The aim of this study is to demonstrate that AZM decreases symptom duration in COVID19 patients and diminishes the viral carriage.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated at the CHU Amiens Picardie presenting:
* Age ≥18 years
* Showing symptoms of COVID -19 and a positive RT-PCR by nasopharyngeal swab
* Non-severe patient, outpatient (not hospitalized), without oxygen
* Having signed a consent to participate in the study

Exclusion Criteria:

* Patient with a contraindication to taking azithromycin, namely: Allergy to macrolides, Severe liver failure.
* In combination with medicines containing cisapride, colchicine, ergotamine or dihydroergotamine
* Pregnant, parturient or breastfeeding women.
* Asymptomatic patients
* Patient unable to be compliant with study protocol
* Patient under guardianship or curators, under the protection of justice or private public law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Length of symptom duration (in days) with azithromycin treatment | up to 2 months
  Length of symptom duration (in days) with azithromycin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Lanoix, Pr, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No